CLINICAL TRIAL: NCT06797908
Title: Pediatric Systemic Hypertension Risk Factors, Complications, Management, and Longitudinal Multidisciplinary Follow-up
Brief Title: Systemic Arterial Hypertension in Pediatric Age.
Acronym: IPERTA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IPERTA
Record Dates: First submitted 2024-12-03; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
We decided to conduct this study because hypertension in childhood increases the risk of developing cardiovascular disease (such as heart attack or stroke) in adulthood, beginning to damage important structures and organs, such as blood vessels, heart, and kidneys, from an early age. There is a clear need to identify those at greatest risk of developing hypertension as early as possible and to follow them appropriately.

The main objectives of the study are to describe the causes of hypertension, study the clinical-laboratory features in the patient with hypertension (such as associated symptoms or conditions, or altered blood test values), evaluate the possible involvement of the heart, and describe the overall approach to the patient with hypertension, from diagnosis (i.e., identification of the condition) to treatment.

DETAILED DESCRIPTION:
The presence and identification of systemic arterial hypertension (hypertension, HTN) in pediatric age has become increasingly relevant in recent years as a consequence of the increase in its prevalence, linked to the change in health determinants witnessed since the late 1970s, such as sedentariness and increased overweight.

In view of the epidemiological consistency of HTN in pediatric age with the possible complications and repercussions in later ages as well, and the economic burden of the management of this patient beginning in early life, both European and North American Guidelines for the child and adolescent on the identification of the individual at risk for HTN and his or her behavioral-pharmacological therapeutic management have been published.

The prevalence of HTN is about 3.5%, while that of elevated blood pressure (BP) is between 2.2 and 3.5% depending on the studies and the population considered, highest in overweight and obese subjects, in whom HTN affects up to 25 percent of subjects, with an increasing incidence trend since the 1980s until reaching a plateau in recent years, consensual with that of obesity. These data underscore the existence of a linear correlation between obesity, metabolic syndrome, and increased blood pressure. Other known conditions that increase the risk of HTN occurrence are prematurity, type 1 diabetes, nephro-vascular and renal diseases with chronic nephropathy, and sleep disorders. Guidance on the definition, diagnosis, and management is provided not only for pathological hypertension but also for high blood pressure values: it has, in fact, been shown that even blood pressure values that are not frankly pathological but nonetheless high can cause organ damage and tend to increase and become pathological within 2 years if left untreated.Longitudinal study cohorts initiated in the 1970s-1980s in both Europe (Young Finns Study) and North America (Framingham Heart Study, Bogalusa Heart Study) have shown that hypertension and cardiovascular (CV) risk factors already present in pediatric age increase CV morbidity and mortality in adults as in a progression of the march of disease. Considering the cardiovascular risk both in the short and long term to which a child diagnosed with systemic hypertension or with normal-to-high blood pressure values is exposed, and the interdependence with metabolic syndrome, endocrine and chronic nephrological pathologies, there is a clear need to identify as early as possible those at higher risk of developing HTN and to appropriately follow up those with elevated blood pressure through early and personalized multidisciplinary interventions. The possibility of recording even longitudinally the evolution of 'possible multidistrict organ damage and its response to treatment could allow us to always modulate therapeutic intervention from the very early stages of the disease and even before the appearance of pathological values. This type of approach would allow us to reduce CV mortality and morbidity even in later ages. The present study is intended to describe the phenomenon of pediatric hypertension with a multidisciplinary approach (cardiovascular, endocrinological and metabolic, and nephrological), with the aim of making the diagnostic-therapeutic-care pathway more effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 18 years of age with hypertension and normal-high blood pressure

Exclusion Criteria:

* Patients with normal blood pressure values

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population will consist of inpatients and outpatients referred to the Center with a diagnosis of hypertension and normal-high blood pressure, according to the European Society of Hypertension Guidelines1
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of diagnostic-therapeutic approach of hypertensionin in a pediatric onset | through study completion, an average of 1 year
  Description of diagnostic-therapeutic approach of hypertensionin in a pediatric onset

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Fabi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Cardiologia Pediatrica e dell'età evolutiva, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve ed Intensiva, Bologna, Bologna
  - IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria, Bologna, Bologna